CLINICAL TRIAL: NCT01365273
Title: Open, Prospective, Randomised Investigation Evaluating Pain With the Use of Mepitel One vs.Bridal Veil and Staples on Split Thickness Skin Grafts
Brief Title: Open, Prosp, Rand. Invest. Evaluating Pain With Mepitel One vs.Bridal Veil and Staples on Split Thickness Skin Grafts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPTO 04
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2012-08

CONDITIONS: Deep Partial Thickness Burn; Full Thickness Burns
Keywords: Split thickness skin grafts; Mepitel One; Bridal Veil and staples; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bridal Veil together with staples (No Intervention): Standard of care. Bridal Veil is fixed over the graft with staples.
- Mepitel One (Active Comparator): Device, dressing
  Interventions: Device: Mepitel One

INTERVENTIONS:
Device: Mepitel One — Dressing
  Arms: Mepitel One

SUMMARY:
This investigation is an open, randomised investigation. Approximately 40 subjects in 4-5 centres in the US with deep-partial of full thickness burns in need of skin grafts will be enrolled.The subjects will be equally randomised to either treatment with Mepitel One or bridal veil together with staples.

The primary objective is to compare pain at the time of dressing change for the use of Mepitel One versus bridal veil together with staples on deep partial or full thickness burns requiring skin grafts.

DETAILED DESCRIPTION:
Skin grafts are placed over excised areas of full thickness injuries and usually attached with sutures or staples. While useful in anchoring the graft in place, subjects often complain of pain from the staples as wound healing progresses.Pulling and sticking are common complaints.There is also a possibility that staples become embedded in the graft which leads to disruption of otherwise healed area, increased pain and anxiety for the subject as well as anxiety for the staff.

Graft take can be optimized with appropriate medical management. Use of non-adherent dressings to protect the graft is customary. Various types of netting-style are used, such as Bridal veil, a sterile product which is fixed over the graft with staples.

Silicone net dressings have also been used successfully to prevent lifting and adherence of skin grafts to the dressings, prevent pain and promote healing. Mepitel One is a sterile, transparent, and flexible wound contact layer consisting of perforated polyurethane film coated with Safetac soft silicone adhesive on one side. Mepitel One is available in various sizes and can be left in place for several days depending on the wound/skin condition.

Evaluation of burns will be performed at Baseline. Skin graft assessment will be performed at Day 7 and Day 14. End of study will be considered the time that graft is considered to have >95% take.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Subjects presenting with 1% - 25% Total Body Surface Area (TBSA) deep partial or full-thickness burns requiring skin graft
  2. At least 1%-10% TBSA is available for grafting that can be considered for study site selection (must have intact, healthy peri-wound area around entire portion of this burned site)
  3. Both genders with age ≥18 years but < 70 years
  4. Signed informed consent

Exclusion Criteria:

1. Subjects with chronic wounds
2. Subjects who are on mechanical ventilation
3. Subjects with dermatologic skin conditions or necrotizing disorders
4. Diagnosed underlying disease(s) (HIV/AIDS, cancer and severe anaemia)judged by the investigator to be a potential interference in the treatment
5. Subjects treated with systemic glucocorticosteroids, except subjects taking occasional doses or doses less than 10 mg prednisolon/day or equivalent
6. Use of immunosuppressive agents, radiation or chemotherapy within the past 30 days
7. Known allergy/hypersensitivity to any of the components of the investigational products
8. Subjects with physical and/or mental conditions that are not expected to comply with the investigation
9. Participation in other clinical investigation(s) within 1 month prior to start of the investigation
10. Previously randomised to this investigation
11. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Patton, MD, Principal Investigator — Nathan Speare Regional Burn Treatment Ctr. Croer Chester Medical Center
Locations (4):
- United States (4):
  - University Foundation for Education & Research, Inc, Tampa, Florida
  - Joseph M. Still Research Foundation, Inc., Augusta, Georgia
  - 5028 Delp Bldg, Mail stop 1011, Kansas City, Kansas
  - Natham Speare Regional Burn Treatment Ctr., Crozer Chester Medical Center, Upland, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first patient included: 26 April 2011 Date of last patient completed: 01 December 2011
Groups:
- Bridal Veil and Staples: Bridal Veil and staples are standard of care I
- Mepitel One: Device
Period: Overall Study
Arm/Group | Bridal Veil and Staples | Mepitel One
Started | 22 | 21
Compl. Pts, Not Evaluable for Pain. | 2 | 4
Completed | 20 | 20
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bridal Veil and Staples | Mepitel One | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (16.0) | 38.0 (18.0) | 40.15 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: VAS Score for Pain Before Dressing Removal
Description: Pain was measured with Visual Analogue Scale (VAS)(100 mm) measuring from 0 = "no pain" at one end to 100 = "most intense pain imagaginable" at the other end.
Time Frame: At visit 6, day 7
Population: All subjects to post-randomization treatment and that provided some data for the primary endpoint were included in the ITT analysis.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Bridal Veil and Staples | Mepitel One
Number analyzed (Participants) | 20 | 17
units on a scale | 11.0 (21.0) | 4.0 (20.1)

2. Primary Outcome: VAS Score for Pain During Dressing Removal
Description: Pain when half of the study product(s) has been removed measued with Visual Analogue Scale (VAS).0 = "no pain" till 100 = "worst pain".
Time Frame: Visit 6, day 7
Population: All included subjects to post-randomization treatment and that provided some data for the primary endpoint was included in the Intention To Treat analyses.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Bridal Veil and Staples | Mepitel One
Number analyzed (Participants) | 20 | 17
units on a scale | 44.0 (28.6) | 4.0 (21.4)

3. Primary Outcome: VAS Score for Pain After Dressing Removal
Description: Pain after the dressing removal measued with Visual Analogue Scale (VAS).0 = "no pain" till 100 = "worst pain".
Time Frame: Visit 6, day 7
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Bridal Veil and Staples | Mepitel One
Number analyzed (Participants) | 20 | 17
units on a scale | 21.0 (34.7) | 3.0 (21.1)

ADVERSE EVENTS:
Arm/Group | Bridal Veil and Staples | Mepitel One
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor is the owner of the results.